CLINICAL TRIAL: NCT01633593
Title: Treatment of Delirium in the Elderly With Donepezil: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects for the trial.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mario R. Louza, MD, PhD, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: deliriumBR2012; 2010/10810-1 (Other Grant/Funding Number: Fapesp); Pfizer (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Elderly; Delirium of Unknown (Axis III) Etiology; Intensive Care (ICU) Myopathy
MeSH Terms: conditions — Muscular Diseases | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- donepezil (Experimental): Donepezil 5mg/day during 2 weeks
  Interventions: Drug: Donepezil
- placebo (Placebo Comparator): placebo comparator to donepezil (double blind)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 5 mg PO a day, during 2 weeks

SUMMARY:
Nowadays features for the diagnosis of delirium are:

1. Disturbance of consciousness (i.e. reduced clarity of environment awareness) with reduced ability to focus, sustain or shift attention;
2. A change in cognition (such as memory deficit, disorientation, language disturbance) or the development of a perceptual disturbance that is not better accounted for by a pre-existing or evolving dementia;
3. The disturbance develops over a short period of time (usually hours to days) and its severity fluctuates during the course of the day;
4. There is evidence from the history, physical examination, or laboratory findings that the disorder is caused by the direct physiological consequences of a general medical condition, substance intoxication or substance withdrawal.

Treatment of underlying clinical disease is important to remit the delirium. However, these procedures alone are not enough to remit the delirium early and to prevent sequels. There is a need for a specific and faster strategy to treat the delirium.

The investigators want to test the hypothesis that an Anticholinesterase Inhibitor (donepezil) can reduce the duration of the delirium.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 year old
* Delirium according to the CAM-ICU (Confusion Assessment Method for Intensive Care Unit)
* informed consent (legal representatives)

Exclusion Criteria:

* unable to swallow pills
* previous allergy to donepezil
* Atrioventricular block of 2nd and 3nd degree

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
reduction of the duration of delirium in elderly patients treated with donepezil | 2 weeks

SECONDARY OUTCOMES:
Severity of delirium (as measured by the DSR-98-R) may influence the response to donepezil | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mario R Louza, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- FAMEMA, Marília, São Paulo, Brazil